CLINICAL TRIAL: NCT00917124
Title: Influence of Intraoperative Monitoring of Cerebral Oximetry on Neurocognitive Function After Coronary Artery Bypass Surgery: Randomized, Prospective Study
Brief Title: Cerebral Oximetry and Neurocognitive Functions in Cardiosurgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Zeljko Colak, Influence of Intraoperative Monitoring of Cerebral Oximetry on Neurocognitive Function After Coronary Artery Bypass Surgery: Randomized, Prospective Study, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KAI-AKA01
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Results first posted 2013-08-07 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: Coronary Artery Disease; Postoperative Cognitive Dysfunction; Neurological Impairment
Keywords: cerebral oximetry; NIRS; INVOS
MeSH Terms: conditions — Coronary Artery Disease; Postoperative Cognitive Complications; Neurologic Manifestations | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- INVOS (Active Comparator): INVOS : Cerebral oxygenation (rSO2) monitoring with INVOS. If rSO2 decreased for more than 20% from patient's baseline value, simple interventions were performed to prevent brain injury. These interventions included: repositioning of head or perfusion cannulae, increasing arterial carbon dioxide tension, increasing oxygen inspiration concentration, increasing arterial blood pressure, adjusting pump flow rate, temperature decreasing, increasing of anesthetic depth and blood transfusion.
  Interventions: Device: INVOS
- CONTROL (No Intervention): The CONTROL arm did not have INVOS or any other cerebral oxygenation monitoring, so interventions to control cerebral oxygenation were not performed.

INTERVENTIONS:
Device: INVOS — Monitoring cerebral oxygenation (rSO2) with INVOS. When rSO2 decline occur it can be responded with simple interventions to prevent a brain injury including: repositioning of the head or perfusion cannulae to avoid mechanical obstruction of cerebral blood flow, increasing arterial carbon dioxide tension within normal referent values, increasing oxygen inspiration concentration to maintain adequate tissue oxygen saturation, increasing arterial blood pressure, pump flow rate and cardiac index, temperature decreasing and increasing of anesthetic depth to reduce cerebral oxygen consumption and blood transfusion if hematocrit decreases below 22%.
  None of the interventions are outside the range of good clinical practice.
  Other Names: INVOS (in vivo optical spectroscopy); NIRS (near infrared spectroscopy)
  Arms: INVOS

SUMMARY:
It is previously reported that the cerebral oxygen desaturation during cardiac surgery is associated with an increased incidence of cognitive impairment. The aim of this study is to determine whether intraoperative monitoring and predetermined interventions protocol to improve cerebral oxygenation during coronary artery bypass surgery provides benefits in neurocognitive functions.

DETAILED DESCRIPTION:
Neurologic complications are major cause of morbidity following coronary artery bypass graft surgery.

The neurologic injuries range in severity from subclinical cognitive changes to fatal brain injury and death. These complications represent a big impact on overall morbidity, and mortality in association with increased costs and length of hospital stay. The social impact is also very important with consequences on patients' quality of life. Several studies reported the incidence of cognitive decline after cardiac surgery that ranges from 30 to 80%. The most common etiologies are embolization and hypoperfusion of the brain.

The In Vivo Optical Spectroscopy (INVOS) system uses near-infrared spectroscopy (NIRS) and provides noninvasive and continuous information on changes in regional oxygen saturation of blood in the brain (rSO2). When rSO2 decline occurs it can be responded with simple interventions to prevent a brain injury. These interventions include: repositioning of the head or perfusion cannulae, increasing arterial carbon dioxide tension, increasing oxygen inspiration concentration, increasing arterial blood pressure, adjusting pump flow rate, temperature decreasing, increasing of anesthetic depth and blood transfusion.

Recent studies reported that intraoperative cerebral oxygen desaturation is associated with early postoperative neuropsychological dysfunction in patients undergoing cardiac surgery.

Neurocognitive function can be assessed with battery of standardized neurocognitive tests. Mini Mental State Examination, Color Trail Test, Grooved Pegboard Test are easy to perform bedside tests that test orientation, registration, attention, calculation, recall, language and complex visual-motor coordination.

ELIGIBILITY:
Inclusion Criteria:

* All patients with coronary artery disease undergoing coronary artery bypass grafting (CABG) with cardiopulmonary bypass

Exclusion Criteria:

* Who refuse to participate
* Previous stroke
* Preexisting psychiatric disease
* Significant carotid stenosis
* Ejection fraction below 25%
* Reoperations
* Emergent surgery
* Dialysis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeljko Colak, MD, Principal Investigator — Clinical Hospital Centre Zagreb
Locations (1):
- University Hospital Center Zagreb, Zagreb, Croatia

REFERENCES:
- [Background] Colak Z, Borojevic M, Bogovic A, Ivancan V, Biocina B, Majeric-Kogler V. Influence of intraoperative cerebral oximetry monitoring on neurocognitive function after coronary artery bypass surgery: a randomized, prospective study. Eur J Cardiothorac Surg. 2015 Mar;47(3):447-54. doi: 10.1093/ejcts/ezu193. Epub 2014 May 7. PMID 24810757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Assessed for eligibility (n=287) Excluded (n=87)
  * Not meeting inclusion criteria (n=79)
  * Declined to participate (n=8)
Groups:
- INVOS: INVOS (In Vivo optical Spectroscopy): Monitoring cerebral oxygenation (rSO2) with INVOS device. When rSO2 decline occur (decrease of rSO2 for more than 20% from patient's baseline value) it can be responded with simple interventions to prevent a brain injury. These interventions include: repositioning of the head or perfusion cannulae, increasing arterial carbon dioxide tension, increasing oxygen inspiration concentration, increasing arterial blood pressure, adjusting pump flow rate, temperature decreasing, increasing of anesthetic depth and blood transfusion.
Period: Overall Study
Arm/Group | CONTROL | INVOS
Started | 100 | 100
Completed | 96 | 94
Not Completed | 4 | 6
Not completed — Protocol Violation | 4 | 6

BASELINE CHARACTERISTICS:
Population: Only patients underwent coronary artery bypass grafting (CABG) with cardiopulmonary bypass were included in the study.
  Four participants in Control group and six participants in INVOS group were not analysed because they did not receive allocated surgical intervention (CABG), because intraoperative plan was changed.
Groups:
- INVOS: INVOS (In Vivo Optical Spectroscopy): Cerebral oxygenation (rSO2) monitoring with INVOS device. If rSO2 decreased for more than 20% from patient's baseline value, simple interventions were performed to prevent brain injury. These interventions included: repositioning of head or perfusion cannulae, increasing arterial carbon dioxide tension, increasing oxygen inspiration concentration, increasing arterial blood pressure, adjusting pump flow rate, temperature decreasing, increasing of anesthetic depth and blood transfusion.
- Total: Total of all reporting groups
Arm/Group | CONTROL | INVOS | Total
Number analyzed (Participants) | 96 | 94 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 64 | 112
  >=65 years | 48 | 30 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (8.8) | 61.9 (7.1) | 62.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 73 | 75 | 148
Region of Enrollment [Number; unit: participants]
  Croatia | 96 | 94 | 190
EuroSCORE [Mean (Standard Deviation); unit: % - predicted mortality] — EuroSCORE (European system for cardiac operative risk evaluation) is a method of calculating predicted operative mortality for patients undergoing cardiac surgery. The outcome (survival or death) was related to the preoperative risk factors. If a risk factor is present in a patient, the weights are added to give an approximate percent predicted mortality. Two online risk calculators are available: the simple additive EuroSCORE and the logistic EuroSCORE. We used the logistic version of EuroSCORE which provides more accurate predicted mortality according to the logistic regression equation.
  % - predicted mortality | 2.4 (1.7) | 2.2 (1.7) | 2.3 (1.7)
Ejection fraction [Mean (Standard Deviation); unit: %] | 56 (9.9) | 56 (9.7) | 56 (9.8)
Years of education [Mean (Standard Deviation); unit: years] | 11.2 (3.2) | 11.3 (3.4) | 11.2 (3.3)
Comorbidity - diabetes [Number; unit: participants]
  Diabetes | 33 | 28 | 61
  Without diabetes | 63 | 66 | 129
Comorbidity - hypertension [Number; unit: participants]
  Hypertension | 85 | 79 | 164
  Without hypertension | 11 | 15 | 26
Comorbidity - Myocardial infarction within 1 month before operation [Number; unit: participants]
  With preoperative myocardial infarction | 12 | 8 | 20
  Without preoperative myocardial infarction | 84 | 86 | 170
Comorbidity - Atrial fibrillation before operation [Number; unit: participants]
  Atrial fibrillation | 5 | 4 | 9
  Without atrial fibrillation | 91 | 90 | 181
Bypass time [Mean (Standard Deviation); unit: minutes] | 89 (32) | 91 (31) | 90 (31)
Aortic cross-clamp time [Mean (Standard Deviation); unit: minutes] | 62 (26) | 63 (23) | 63 (25)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Incidence of Cognitive Impairment Between Groups. Change Between Preoperative and Postoperative Cognitive Function Was Assessed by Performing Standardized Neurocognitive Tests.
Description: The Mini-Mental State Examination (MMSE) total score is calculated by summing the item scores across several aspects of cognition. The maximum possible total score is 30 points.
  Color Trials Test (CTT) measures sustained visual attention, visual scanning and graphomotor skills. The examiner records the length of time (in seconds) required by the patient to rapidly draw a line connecting the circles numbered 1 through 25 in consecutive order.
  Grooved-Pegboard test (GP test) is manipulative dexterity test that contains twenty-five holes with randomly positioned slots and pegs which have a key along one side. Pegs must be rotated to match the hole before they can be inserted. The examiner records the time in seconds.
  Cognitive impairment was defined as a decline in postoperative performance in one or more tests: decrease of MMSE score three points or more from baseline and decrease of one standard deviation or more in performance on CTT 1 and GP tests
Time Frame: preoperative, 7 days postoperative
Population: 3 participants in Control group did not perform control cognitive test- transferred to another hospital.
  6 participants in INVOS group did not perform control cognitive test - transferred to another hospital n=4, declined to participate n=2
Measure: Number; unit: participants
Arm/Group | CONTROL | INVOS
Number analyzed (Participants) | 93 | 88
participants | 48 | 25
Statistical Analysis 1: Comparison: CONTROL vs INVOS; Hypothesis: intraoperative monitoring of cerebral oxigenation with INVOS system will improve cognitive outcome of patients undergoing CABG procedure. Sample size was determined assuming 50% incidence of cognitive impairment after cardiac surgery and possibility of decreasing that incidence to 30% using cerebral oximetry. Based on 0.8 power to detect a significant difference (p=0.05), 90 patients were required for each study group; Test type: Superiority or Other; p = 0.002, Chi-squared, Corrected

2. Secondary Outcome: Evidence of Coma, Stupor, Cerebral Insult, Delirium, Ventilation Longer Than 24 Hours, Myocardial Infarction, Atrial Fibrillation, Dialysis, Reoperation for Bleeding, Infection, Hospital Stay > 7 Days
Time Frame: 7 postoperative days
Measure: Number; unit: participants
Arm/Group | CONTROL | INVOS
Number analyzed (Participants) | 96 | 94
participants
  Stroke, coma, stupor | 1 | 4
  Delirium | 13 | 8
  Prolonged mechanical ventilation | 2 | 1
  Myocardial infarction | 7 | 7
  Hemodialysis | 1 | 0
  Infection (any type) | 18 | 17
  Revision for bleeding | 1 | 0
  Atrial fibrillation | 26 | 21
  Hospital stay > 7 days | 43 | 44

ADVERSE EVENTS:
Time Frame: seven postoperative days
Groups:
- INVOS: INVOS : Monitoring cerebral oxygenation (rSO2) with INVOS. When rSO2 decline occur (decrease of rSO2 for more than 20% from patient's baseline value) it can be responded with simple interventions to prevent a brain injury. These interventions include: repositioning of the head or perfusion cannulae, increasing arterial carbon dioxide tension, increasing oxygen inspiration concentration, increasing arterial blood pressure, adjusting pump flow rate, temperature decreasing, increasing of anesthetic depth and blood transfusion.
Arm/Group | INVOS | CONTROL
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/96
Other Adverse Events (participants affected / at risk) | 0/94 | 0/96

LIMITATIONS AND CAVEATS:
* number and selection of performed neurocognitive tests. MMSE test is not part of "Statement of consensus on assessment of neurobehavioral outcomes after cardiac surgery"
* lack of blind monitoring of cerebral oximetry in control group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No